CLINICAL TRIAL: NCT04872010
Title: Construction of a Database for the Life-cycle Sepsis-specific Disease Cohort
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Shuming Pan, Deputy Dean of Xinhua Hospital, Leader of Emergency Medicine Science Department, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHDC2020CR6030
Record Dates: First submitted 2021-04-10; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establish a structured clinical database for sepsis screening, and establish a special data set standard for sepsis throughout the life cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sepsis who meet the Sepsis 3.0 standard proposed by the 2016 International Sepsis Expert Consensus, that is, for patients with infection or suspected infection, when sepsis-related sequential organ failure (Sequential (Sepsis-related) Organ Failure) Assessment (SOFA) score increased by ≥ 2 points from the baseline can be diagnosed as sepsis;
2. It is estimated that the patient's ICU stay ≥24 hours;
3. Obtain informed consent and sign an informed consent form.

Exclusion Criteria:

1. The patient's ICU hospital stay is less than 24 hours;
2. Participated in other clinical research;
3. Failed to sign the informed consent form.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1-100 years
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Sepsis organ function status and survival analysis. | 2022.09.30
  Safety indicators include: prognosis: mortality, intensive care unit (ICU) treatment time and hospital stay, incidence of nosocomial infections, treatment-related complications.

IPD SHARING:
Plan to Share IPD: No